CLINICAL TRIAL: NCT00004451
Title: Randomized Study of the Effects of Glucose on Cognition in Healthy Young and Elderly People and Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: University of Virginia (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13548; K07MH001197 (NIH)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Glucose

INTERVENTIONS:
Drug: Glucose

SUMMARY:
This study will determine whether glucose facilitates memory in healthy elderly people and those with Parkinson's disease.

DETAILED DESCRIPTION:
Subjects fast for 8 hours before receiving a test to determine their blood glucose levels. Following this test, subjects are randomized to receive either a glucose or saccharin sweetened drink. A series of memory tests and an additional 3 blood glucose level tests are administered approximately 15 minutes later. A minimum of 1 week afterward, the subjects return and receive the alternate sweetener followed by additional memory tests.

ELIGIBILITY:
Inclusion Criteria:

* Three groups of subjects are eligible for this study: Healthy young adults between ages 18 and 30; Healthy elderly adults between ages 60 and 90; AND Anyone diagnosed with Parkinson's disease

Exclusion Criteria:

* Prior surgery to remove part of the stomach
* Diabetes, Addison's, or Cushing's diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Manning, Study Chair — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States